CLINICAL TRIAL: NCT04551898
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of SARS-CoV-2 Neutralizing Antibody BGB-DXP593 in Patients With Mild-to-Moderate COVID-19
Brief Title: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Neutralizing Antibody BGB-DXP593 in Participants With Mild-to-Moderate Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-DXP593-102
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Results first posted 2022-03-17 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BGB-DXP593 Low Dose (Experimental): Participants will receive BGB-DXP593 on Day 1, and followed up for safety for up to 85 days
  Interventions: Drug: BGB-DXP593
- BGB-DXP593 Medium Dose (Experimental): Participants will receive BGB-DXP593 on Day 1, and followed up for safety for up to 85 days
  Interventions: Drug: BGB-DXP593
- BGB-DXP593 High Dose (Experimental): Participants will receive BGB-DXP593 on Day 1, and followed up for safety for up to 85 days
  Interventions: Drug: BGB-DXP593
- Placebo (Placebo Comparator): Participants will receive placebo on Day 1, and followed up for safety for up to 85 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGB-DXP593 — Intravenous (IV) infusion administered over 30 to 90 minutes at a dose as specified in the treatment arm
  Arms: BGB-DXP593 High Dose; BGB-DXP593 Low Dose; BGB-DXP593 Medium Dose
Drug: Placebo — Placebo to match BGB-DXP593 administered as specified in the treatment arm
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of BGB-DXP593 administered intravenously as a single dose in participants with mild to moderate COVID-19

ELIGIBILITY:
Key Inclusion Criteria:

1. Laboratory-confirmed severe acute respiratory syndrome (SARS)-CoV-2 infection (positive reverse transcription-polymerase chain reaction [RT-PCR] test or other authorized antigen testing methods) in any samples following local practice ≤ 72 hours prior to screening.
2. Have experienced COVID-19 symptoms for ≤ 7 days prior to treatment assignment, such as fever, cough, shortness of breath, sore throat, diarrhea, vomiting, and dysgeusia
3. Agree to the collection of nasopharyngeal swabs, saliva, and venous blood

Key Exclusion Criteria:

1. Severe COVID-19 having oxygen saturation (SpO2) ≤ 93 % on room air at sea level or ratio of arterial oxygen partial pressure (PaO2 in millimeters of mercury) to fractional inspired oxygen (FiO2) < 300, respiratory rate ≥ 30/min, heart rate ≥ 125/min
2. Requires mechanical ventilation or anticipated impending need for mechanical ventilation
3. Known allergies to any of the components used in the formulation of the interventions
4. Have received an investigational intervention for SARS-CoV-2 prophylaxis within 30 days before dosing
5. Have received treatment with a SARS-CoV-2 specific monoclonal antibody

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (18):
- United States (11):
  - Btc Network Midland Florida Clinical Research Center, DeLand, Florida
  - Elixia Clinical Research Collaborative, Hollywood, Florida
  - Homestead Associates in Research Inc, Miami, Florida
  - Medical Research Center of Miami Ii, Inc, Miami, Florida
  - Us Associates in Research, Miami, Florida
  - Continental Research Network, Miami, Florida
  - Orlando Health Ufhealth Cancer Center, Orlando, Florida
  - Revive Research Institute, Dearborn, Michigan
  - Revival Research Institute Farmington Hills, Sterling Heights, Michigan
  - Amarillo Center For Clinical Research, Amarillo, Texas
  - Panamerican Clinical Research Us Headquarters, Brownsville, Texas
- Brazil (3):
  - Hospital Das Clinicas Da Faculdade de Medicina de Botucatu, Botucatu
  - Fundacao Universidade de Caxias Do Sul, Caxias do Sul
  - Consultoria Medica E Pesquisa Clinica, Sorcaba
- Mexico (2):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - IECSI, Monterrey
- South Africa (2):
  - Task Clinical Research Centre, Cape Town
  - Langeberg Clinical Trials, Cape Town

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Vega R, Antila M, Perez C, Mookadam M, Xie F, Zhang W, Rizwan A, Yao Z, Rasko JEJ. SARS-CoV-2-neutralising antibody BGB-DXP593 in mild-to-moderate COVID-19: a multicentre, randomised, double-blind, phase 2 trial. EClinicalMedicine. 2023 Mar;57:101832. doi: 10.1016/j.eclinm.2023.101832. Epub 2023 Feb 16. PMID 36820098
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 20 centers and 181 participants were treated.
Groups:
- Placebo: Single intravenous infusion of placebo solution administered over 30 to 90 minutes
- BGB-DXP593 5 mg/kg: Single intravenous infusion of 5 milligrams/kilogram (mg/kg) DXP593 administered for 30 to 90 minutes
- BGB-DXP593 15 mg/kg: Single intravenous infusion of 15 mg/kg DXP593 administered for 30 to 90 minutes
- BGB-DXP593 30 mg/kg: Single intravenous infusion of 30 mg/kg DXP593 administered for 30 to 90 minutes
Period: Overall Study
Arm/Group | Placebo | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Started | 47 | 45 | 43 | 46
Completed | 39 | 42 | 35 | 41
Not Completed | 8 | 3 | 8 | 5
Not completed — Participant randomized but did not receive study drug | 0 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 2 | 2
Not completed — Lost to Follow-up | 2 | 1 | 2 | 2
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Incorrectly randomized and screen failed due to administrative error | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set includes all randomized participants.
Groups:
- BGB-DXP593 5 mg/kg: Single intravenous infusion of 5 mg/kg DXP593 administered over 30 to 90 minutes
- BGB-DXP593 15 mg/kg: Single intravenous infusion of 15 mg/kg DXP593 administered over 30 to 90 minutes
- BGB-DXP593 30 mg/kg: Single intravenous infusion of 30 mg/kg DXP593 administered over 30 to 90 minutes
- Total: Total of all reporting groups
Arm/Group | Placebo | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg | Total
Number analyzed (Participants) | 47 | 45 | 43 | 46 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (14.02) | 46.2 (15.56) | 43.6 (12.43) | 41.1 (13.35) | 43.8 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 22 | 27 | 86
  Male | 27 | 28 | 21 | 19 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 1 | 2 | 8
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 2 | 5 | 15
  White | 40 | 35 | 39 | 33 | 147
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 8 in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Viral Shedding
Description: SARS-CoV-2 viral shedding was measured by reverse transcription-quantitative polymerase chain reaction (RT-qPCR) in nasopharyngeal swab samples.
Time Frame: Baseline and Day 8
Population: Intent To Treat (ITT) analysis set. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: log10 copies/ml
Arm/Group | Placebo | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 41 | 42 | 34 | 42
log10 copies/ml | -2.88 (2.241) | -3.52 (2.831) | -3.75 (2.513) | -3.03 (2.239)
Statistical Analysis 1: Comparison: Placebo vs BGB-DXP593 5 mg/kg; Test type: Superiority; p = 0.4829, Mixed Models Analysis; Least square Mean = -0.25, 90% CI 2-sided [-0.84 to 0.34]
Statistical Analysis 2: Comparison: Placebo vs BGB-DXP593 15 mg/kg; Test type: Superiority; p = 0.1739, Mixed Models Analysis; Least square Mean = -0.51, 90% CI 2-sided [-1.13 to 0.11]
Statistical Analysis 3: Comparison: Placebo vs BGB-DXP593 30 mg/kg; Test type: Superiority; p = 0.6006, Mixed Models Analysis; Least square Mean = 0.19, 90% CI 2-sided [-0.40 to 0.77]
Statistical Analysis 4: Comparison: Placebo vs BGB-DXP593 5 mg/kg vs BGB-DXP593 15 mg/kg vs BGB-DXP593 30 mg/kg; Test type: Superiority; p = 0.4996, t-test, 1 sided — H0: there is a flat dose response curve comparing change from baseline to Day 8 in viral load in the Placebo and other BGB-DXP593 dose groups; MCP Mod was used to test the primary hypothesis and provide 1-sided p-value accordingly

2. Secondary Outcome: Time-Weighted Average Change in SARS-CoV-2 Viral Shedding From Baseline to Day 15
Time Frame: Baseline and Day 15
Population: ITT analysis set. Participants with available samples were included in the analysis.
Measure: Mean (Standard Deviation); unit: log10 copies/ml
Arm/Group | Placebo | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 45 | 43 | 37 | 44
log10 copies/ml | -2.56 (1.718) | -2.93 (1.997) | -2.87 (2.049) | -2.55 (1.785)

3. Secondary Outcome: Change in SARS-CoV-2 Viral Shedding From Baseline to Day 15
Description: SARS-CoV-2 viral shedding was measured by RT-qPCR in nasopharyngeal swab samples
Time Frame: Baseline and Day 15
Population: ITT analysis set. Participants with available samples were included in the analysis.
Measure: Mean (Standard Deviation); unit: log10 copies/ml
Arm/Group | Placebo | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 41 | 41 | 32 | 42
log10 copies/ml | -4.16 (2.446) | -4.29 (2.675) | -4.31 (2.851) | -4.04 (2.577)

4. Secondary Outcome: Time to Negative RT-qPCR in All Tested Samples
Description: The negative RT-qPCR is defined as the value that is below the lower limit of detection
Time Frame: From Baseline up to Day 21
Population: ITT analysis set
Measure: Median (90% Confidence Interval); unit: Days
Groups:
- BGB-DXP593 5 mg/kg: Single intravenous infusion of 5 mg/kg DXP593 administered for 30 to 90 minutes
Arm/Group | Placebo | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 47 | 45 | 43 | 46
Days | 17.00 [15.00 to 19.00] | 15.00 [13.00 to 17.00] | 10.00 [8.00 to 16.00] | 17.00 [15.00 to 17.00]

5. Secondary Outcome: Percentage of Participants Who Required Hospitalization Due to Worsened COVID-19
Time Frame: Baseline up to End of Study (EOS) /174 Days
Population: ITT analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 47 | 45 | 43 | 46
Percentage of participants | 4.3 | 2.2 | 2.3 | 0.0

6. Secondary Outcome: Time to Resolution of All COVID-19-Related Symptoms
Time Frame: Baseline up to EOS /174 Days
Population: ITT analysis set
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Placebo | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 47 | 45 | 43 | 46
Days | 16.5 [14.00 to 22.00] | 15.0 [14.00 to 22.00] | 19.0 [15.00 to 22.00] | 14.0 [9.00 to 16.00]

7. Secondary Outcome: All-Cause Mortality at Day 29
Description: Number of participants that died by Day 29
Time Frame: Day 29
Population: ITT analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 47 | 45 | 43 | 46
Percentage of participants | 2.13 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Up to 174 days
Population: Safety analysis set includes all participants who received the study drug or placebo.
Measure: Number; unit: Number of participants
Arm/Group | Placebo | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 47 | 44 | 40 | 45
Number of participants
  With at Least One TEAE | 6 | 6 | 4 | 7
  Grade 3 or Higher TEAE | 1 | 1 | 1 | 0
  Serious TEAE | 2 | 2 | 1 | 0

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of BGB-DXP593
Time Frame: Day 1 (pre-dose, End of Infusion) Days 3, 8, 15, 29, and End of study visit (up to174 days)
Population: Pharmacokinetic (PK) analysis set includes all participants who have received the study drug per protocol and for whom PK data are available.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 42 | 40 | 44
µg/mL | 132.95 (53.180) | 368.22 (232.040) | 714.17 (149.198)

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) of BGB-DXP593 From Time 0 to Day 29
Time Frame: Day 1 (pre-dose, End of Infusion) Days 3, 8, 15, and 29
Population: PK analysis set includes all participants who have received the study drug per protocol and for whom PK data are available.
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 42 | 37 | 45
day*μg/mL | 1188.7 [620 to 3540] | 3014.3 [1198 to 4159] | 6609.2 [4345 to 8989]

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) of BGB-DXP593
Description: AUClast : AUC from time zero to the time of the last quantifiable concentration AUCinf: AUC from zero to infinite time with extrapolation of the terminal phase
Time Frame: Day 1 (pre-dose, End of Infusion) Days 3, 8, 15, 29, and End of study visit (up to 174 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 43 | 40 | 45
day*μg/mL
  AUClast | 1829.3 [843 to 4491] | 4707.5 [406 to 6883] | 10259.5 [5165 to 16198]
  AUCInf: number analyzed (Participants) | 38 | 35 | 40
  AUCInf | 2098.7 [851 to 4564] | 4996.3 [2065 to 7351] | 10509.2 [5816 to 17245]

12. Secondary Outcome: Time to Reach Cmax (Tmax) of BGB-DXP593
Time Frame: Day 1 (pre-dose, End of Infusion) Days 3, 8, 15, 29, and End of study visit (up to 174 days)
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 43 | 40 | 45
hours | 1.500 [0.75 to 322.72] | 1.500 [0.73 to 35.50] | 1.500 [0.83 to 34.25]

13. Secondary Outcome: Terminal Half-Life (t1/2) of BGB-DXP593
Time Frame: Day 1 (pre-dose, End of Infusion) Days 3, 8, 15, 29, and End of study visit (up to 174 days)
Population: as for outcome 9
Measure: Median (Full Range); unit: Day
Arm/Group | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 38 | 35 | 40
Day | 21.4 [15 to 40] | 23.2 [15 to 32] | 20.8 [14 to 32]

14. Secondary Outcome: Clearance (CL) of BGB-DXP593
Time Frame: Day 1 (pre-dose, End of Infusion) Days 3, 8, 15, 29, and End of study visit (up to 174 days)
Population: as for outcome 9
Measure: Median (Full Range); unit: Liters/Day
Arm/Group | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 38 | 35 | 40
Liters/Day | 0.21 [0.1 to 0.5] | 0.25 [0.2 to 0.5] | 0.24 [0.1 to 0.4]

15. Secondary Outcome: Volume of Distribution During the Terminal Phase (Vz) of BGB-DXP593
Time Frame: Day 1 (pre-dose, End of Infusion) Days 3, 8, 15, 29, and End of study visit (up to 174 days)
Population: as for outcome 9
Measure: Median (Full Range); unit: Liters
Arm/Group | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 38 | 35 | 40
Liters | 6.58 [2.5 to 11.9] | 8.07 [5.2 to 18.9] | 7.33 [3.3 to 11.6]

16. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs) to BGB-DXP593
Time Frame: Day 1 (pre-dose) Days 15, 29, and End of study visit (up to 174 days)
Population: The ADA Analysis Set includes all the participants who have received the study drug and in whom both baseline ADA and at least 1 postbaseline ADA results are available
Measure: Number; unit: Number of participants
Arm/Group | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 44 | 37 | 45
Number of participants
  Treatment Induced | 1 | 0 | 0
  Neutralizing antibody Positive | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 174 days
Description: Safety Analysis Set included all participants who received the study drug or placebo.
Arm/Group | Placebo | BGB-DXP593 5 mg/kg | BGB-DXP593 15 mg/kg | BGB-DXP593 30 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/47 | 0/44 | 0/40 | 0/45
Serious Adverse Events (participants affected / at risk) | 2/47 | 2/44 | 1/40 | 0/45
Other Adverse Events (participants affected / at risk) | 5/47 | 4/44 | 4/40 | 7/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | BGB-DXP593 5 mg/kg (N=44) | BGB-DXP593 15 mg/kg (N=40) | BGB-DXP593 30 mg/kg (N=45)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | BGB-DXP593 5 mg/kg (N=44) | BGB-DXP593 15 mg/kg (N=40) | BGB-DXP593 30 mg/kg (N=45)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site hypersensitivity (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT04551898/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT04551898/SAP_001.pdf